CLINICAL TRIAL: NCT00854230
Title: Pharmacotherapy for HIV Infected Patients With Alcohol Problems
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We expanded to a bigger, multi-site study & decided to close this study.
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJ0007; 0901004647
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infection; Heavy Alcoholic Consumption; HIV Infections
Keywords: HIV; alcohol; naltrexone; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Naltrexone
  Interventions: Drug: Naltrexone
- 2 (Placebo Comparator)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltrexone dose 25-100mg
  Other Names: Revia

SUMMARY:
This is a randomized double blind clinical trial to test the effect of Naltrexone on HIV infected heavy drinkers. The study will select 40 HIV positive patients who meet criteria for heavy drinking. Treatments include Naltrexone (25-100mg)and placebo. Patients will be treated, followed up, and assessed for a duration of 12 weeks.

The investigators associated hypotheses Hypothesis 1: Naltrexone will reduce the frequency of heavy drinking. Hypothesis 2: Naltrexone will lead to maintenance or improvement in CD4 lymphocyte count and decreased HIV RNA levels.

Hypothesis 3: Naltrexone will lead to a reduction in sexual risk behaviors. Hypothesis 4: Naltrexone will lead to improved adherence to HAART. Hypothesis 5 (Exploratory): Naltrexone will be well-tolerated with minimal side effects and patients will exhibit good treatment retention.

ELIGIBILITY:
Inclusion Criteria:

1. Be HIV-positive.
2. Report heavy drinking 4 or more times in the past 4 weeks. Heavy drinking is defined as 4 or more drinks for women and 5 or more drinks for men on any occasion.
3. Not be abstinent from alcohol for greater than 30 days.
4. Be at least 18 years old.
5. Be able to understand English and provide informed consent

Exclusion Criteria:

1. Be psychotic or severely psychiatrically disabled.
2. Have medical conditions that would preclude completing or be of harm during the course of the study.
3. Have laboratory or clinical evidence of significant liver dysfunction (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of the normal range) or cirrhosis.
4. Have a known contraindication to naltrexone therapy (e.g. taking opioid medication for pain).
5. Be pregnant, nursing or unable to use an effective method of birth control (women).
6. Subjects who are taking or use narcotics will not be included because naltrexone will precipitate withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Frequency of heavy drinking | 12 weeks

SECONDARY OUTCOMES:
HIV biological markers | 12 weeks
Sexual risk behavior | 12 weeks
Tolerability and retention in alcohol treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David A Fiellin, Md, Principal Investigator — Yale University; Amy Justice, MD, PhD, Principal Investigator — Yale University, West Haven VA hospital